CLINICAL TRIAL: NCT02993614
Title: Characteristics and Cardiovascular and Mortality Outcomes in Patients With Type 2 Diabetes Mellitus Initiating Treatment With Sodium-glucose Co-transporter-2 Inhibitors (SGLT-2i) and Other Glucose Lowering Drugs
Brief Title: Comparative Effectiveness of Cardiovascular Outcomes in New Users of SGLT-2 Inhibitors
Acronym: CVD-REAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00015
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
CVD-REAL is a multinational, observational cohort study in patients with type 2 diabetes mellitus evaluating the comparative effectiveness of initiating treatment with a sodium-glucose co-transporter-2 (SGLT-2) inhibitor versus another glucose-lowering drug. This study will compare the risk of all-cause mortality and clinically relevant cardiovascular (CV) outcomes respectively in patients who are new users of SGLT-2 inhibitors with those who are new users of other glucose-lowering drugs. CVD-REAL is aiming to collect data from approximately 4 million patients overall, from twelve countries across three major world regions.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus remains a major risk factor for cardiovascular disease with an estimated 425 million adults worldwide having diabetes in 2017, with type 2 diabetes mellitus accounting for about 90% of the cases. Recent evidence indicates that certain glucose-lowering therapies are associated with reduction in cardiovascular outcomes. There is, therefore, an urgent need to improve the understanding of the impact of newer classes of glucose-lowering therapies, such as dipeptidyl peptidase-4 (DPP-4) inhibitors, glucagon-like peptide-1 (GLP-1) receptor agonists and sodium-glucose co-transporter-2 (SGLT-2) inhibitors on cardiovascular outcomes in clinical practice.

CVD-REAL is a comparative effectiveness study that aims to compare new users of SGLT-2 inhibitors with new users of other glucose-lowering drugs with regard to the risk of all-cause mortality and clinically relevant CV outcomes (including stroke, myocardial infarction, and hospitalization for heart failure) respectively. The study is based on data from 12 countries across four major world regions.

The study is conducted using data from claims, medical records and national health registries from twelve countries combined in two waves. CVD-REAL 1 includes Germany, Denmark, Norway, Sweden, United Kingdom (UK) and United States of America (USA). CVD-REAL 2 comprises Australia, Canada, Israel, Japan, Singapore and South Korea. The study will collect data from approximately 4 million patients from the time they start treatment with a SGLT-2 inhibitor or another glucose-lowering drug (index date) to the end of the follow-up period.

The Study Population will consist of new users of SGLT-2i and other glucose lowering drugs respectively. These will be compared with all-cause mortality, hospitalization for heart failure, myocardial infarction and stroke during the follow-up period. In addition certain other cardiovascular and renal outcomes will be assessed descriptively in the two groups respectively.

The study period will range from launch of the first SGLT-2i in each of the countries and end at latest available data in each data source.

All-cause mortality and the incidence of cardiovascular events will be compared between new users of SGLT-2 inhibitors and the comparator arm using a hazard ratio (relative risk) and corresponding 95% confidence interval. The analysis will be performed using the Cox proportional hazards model or some other appropriate method.

Matching by propensity scores will be used to balance the potential confounding covariates between the SGLT-2i group and the reference group to ensure that the two groups are as similar as possible at baseline.To achieve sufficient power, a meta-analysis will be applied to integrate the point estimates from each of the individual database analyses and calculate an overall weighted estimate and corresponding 95% CI.

ELIGIBILITY:
Inclusion Criteria:

* New user receiving or dispensed prescription of SGLT-2i medication or other glucose lowering drug, oral as well as injectable, including fixed-dose combination (FDC) products containing these medication groups
* T2DM diagnosis on or prior to the index date
* ≥ 18 years old at index date
* > 1 year data history in the database prior to the index date

Exclusion Criteria:

* Patients with a T1DM diagnosis
* Patients with gestational diabetes within 1 year before index date

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New users of SGLT--2i and other glucose lowering drugs respectively
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
CVD REAL1 Incidence of hospitalization for heart failure. / CVD REAL 2 All-cause mortality | From index date up to latest available data of first prescription of an SGLT-2i or a new oGLD in each of the countries ranging from Sep 11 (UK) until Apr 15 (IL) until the last date of data collection or outcome ranging from Sep 15 (US) to Nov 17 (SG)
  Heart failure events obtained from general practice or hospital records, electronic health records or national health registers; All-cause mortality obtained from linkeage to death national registers

SECONDARY OUTCOMES:
CVD REAL1 All-cause mortality; CVD REAL 2: Hospitalization for heart failure (HHF), stroke, myocardial infarction (MI) and including composite endpoints | From index date up to latest available data of first prescription of an SGLT-2i or a new oGLD in each of the countries ranging from Sep 11 (UK) until Apr 15 (IL) until the last date of data collection or outcome ranging from Sep 15 (US) to Nov 17 (SG)
  Events obtained from general practice or hospital records, electronic health records and national health registers. All cause mortality obtained from linkeage to death national registers

CONTACTS AND LOCATIONS:
Locations (17):
- Research Site, Wilmington, Delaware, United States
- Research Site, Melbourne, D1690r00015, Australia
- Research Site, Mississauga, D1690r00015, Canada
- Research Site, Gentofte Municipality, D1690r00015, Denmark
- Research Site, Espoo, D1690r00015, Finland
- Research Site, Ulm, D1690r00015, Germany
- Research Site, Raanana, D1690r00015, Israel
- Research Site, Rome, D1690r00015, Italy
- Research Site, Tokyo, D1690r00015, Japan
- Research Site, Oslo, D1690r00015, Norway
- Research Site, Porto, D1690r00015, Portugal
- Research Site, Singapore, D1690r00015, Singapore
- Research Site, Seoul, D1690r00015, South Korea
- Research Site, Madrid, D1690r00015, Spain
- Research Site, Södertälje, D1690r00015, Sweden
- Research Site, Taipei, D1690r00015, Taiwan
- Research Site, Luton, D1690r00015, United Kingdom

REFERENCES:
- [Derived] Khunti K, Kosiborod M, Kim DJ, Kohsaka S, Lam CSP, Goh SY, Chiang CE, Shaw JE, Cavender MA, Tangri N, Franch-Nadal J, Holl RW, Jorgensen ME, Norhammar A, Eriksson JG, Zaccardi F, Karasik A, Magliano DJ, Thuresson M, Chen H, Wittbrodt E, Bodegard J, Surmont F, Fenici P; CVD-REAL Investigators and Study Group. Cardiovascular outcomes with sodium-glucose cotransporter-2 inhibitors vs other glucose-lowering drugs in 13 countries across three continents: analysis of CVD-REAL data. Cardiovasc Diabetol. 2021 Jul 31;20(1):159. doi: 10.1186/s12933-021-01345-z. PMID 34332558
- [Derived] Nicolucci A, Candido R, Cucinotta D, Graziano G, Rocca A, Rossi MC, Tuccinardi F, Manicardi V. Generalizability of Cardiovascular Safety Trials on SGLT2 Inhibitors to the Real World: Implications for Clinical Practice. Adv Ther. 2019 Oct;36(10):2895-2909. doi: 10.1007/s12325-019-01043-z. Epub 2019 Aug 13. PMID 31410779
- [Derived] Cavender MA, Norhammar A, Birkeland KI, Jorgensen ME, Wilding JP, Khunti K, Fu AZ, Bodegard J, Blak BT, Wittbrodt E, Thuresson M, Fenici P, Hammar N, Kosiborod M; CVD-REAL Investigators and Study Group. SGLT-2 Inhibitors and Cardiovascular Risk: An Analysis of CVD-REAL. J Am Coll Cardiol. 2018 Jun 5;71(22):2497-2506. doi: 10.1016/j.jacc.2018.01.085. PMID 29852973
- [Derived] Kosiborod M, Lam CSP, Kohsaka S, Kim DJ, Karasik A, Shaw J, Tangri N, Goh SY, Thuresson M, Chen H, Surmont F, Hammar N, Fenici P; CVD-REAL Investigators and Study Group. Cardiovascular Events Associated With SGLT-2 Inhibitors Versus Other Glucose-Lowering Drugs: The CVD-REAL 2 Study. J Am Coll Cardiol. 2018 Jun 12;71(23):2628-2639. doi: 10.1016/j.jacc.2018.03.009. Epub 2018 Mar 11. PMID 29540325
- [Derived] Kosiborod M, Cavender MA, Fu AZ, Wilding JP, Khunti K, Holl RW, Norhammar A, Birkeland KI, Jorgensen ME, Thuresson M, Arya N, Bodegard J, Hammar N, Fenici P; CVD-REAL Investigators and Study Group*. Lower Risk of Heart Failure and Death in Patients Initiated on Sodium-Glucose Cotransporter-2 Inhibitors Versus Other Glucose-Lowering Drugs: The CVD-REAL Study (Comparative Effectiveness of Cardiovascular Outcomes in New Users of Sodium-Glucose Cotransporter-2 Inhibitors). Circulation. 2017 Jul 18;136(3):249-259. doi: 10.1161/CIRCULATIONAHA.117.029190. Epub 2017 May 18. PMID 28522450
- See also: CSP_D1690R00015. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14609&filename=CSP_D1690R00015.pdf
- See also: CSP_amendment_D1690R00015. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14609&filename=CSP_amendment_D1690R00015.pdf
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690R00015&attachmentIdentifier=8e066078-f806-4731-a5d6-607baa08816f&fileName=CSR_CVD-REAL_15_Dec_redacted.docx&versionIdentifier=